CLINICAL TRIAL: NCT05289050
Title: Analgesic Effect of Intraoperative Intravenous S-Ketamine During Total Knee Arthroplasty Surgery:A Randomized Controlled Clinical Trial
Brief Title: Analgesic Effect of Intraoperative Intravenous S-Ketamine During Total Knee Arthroplasty Surgery
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ling Dong (Other)
Responsible Party: Sponsor-Investigator, Ling Dong, clinical professor, Qianfoshan Hospital
Organization: Qianfoshan Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: YXLL-KY-2021(077)
Record Dates: First submitted 2022-02-26; First posted 2022-03-21 (Actual); Last update posted 2023-02-28 (Actual); Status verified 2023-02

CONDITIONS: Postoperative Pain, Acute; Anaesthetic
Keywords: Postoperative pain; total knee arthroplasty surgery; anaesthetic; S-ketamine infusion
MeSH Terms: conditions — Pain, Postoperative | interventions — Sodium Chloride; Esketamine

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- sodium chloride (NaCl; 0.9%) (Placebo Comparator): For patients in the control group,anaesthesia will be maintained with intravenous sodium chloride (NaCl; 0.9%) infusion.while anaesthesia will be maintained with propofol infusion(4-12mg/kg/h),analgesia will be maintained with remifentanil(0.15-0.3ug/kg/min).The sufentanil dose at induction and the rate of intraoperative remifentanil and propofol infusions were at the discretion of the anesthesiologist in charge of the patient. The assessment of the depth of anesthesia was based on clinical evaluation,placebo-controlled infusion will be stopped 15 minutes before the end of surgery.Propofol and remifentanil infusion will be stopped at the end of surgery.
  Interventions: Drug: sodium chloride (NaCl; 0.9%)
- S-ketamine (Experimental): For patients in the s-ketamine group, anaesthesia will be maintained with s-ketamine infusion（0.3mg/kg/h),while anaesthesia will be maintained with propofol infusion(4-12mg/kg/h) ,analgesia will be maintained with remifentanil(0.15-0.3ug/kg/min).The sufentanil dose at induction and the rate of intraoperative remifentanil and propofol infusions were at the discretion of the anesthesiologist in charge of the patient.The assessment of the depth of anesthesia was based on clinical evaluation.S-ketamine infusion will be stopped 15 minutes before the end of surgery.Propofol and remifentanil infusion will be stopped at the end of surgery.
  Interventions: Drug: S-ketamine

INTERVENTIONS:
Drug: sodium chloride (NaCl; 0.9%) — For patients in the control group,anaesthesia will be maintained with intravenous sodium chloride (NaCl; 0.9%) infusion.while anaesthesia will be maintained with propofol infusion(4-12mg/kg/h),analgesia will be maintained with remifentanil(0.15-0.3ug/kg/min).The sufentanil dose at induction and the rate of intraoperative remifentanil and propofol infusions were at the discretion of the anesthesiologist in charge of the patient.The assessment of the depth of anesthesia was based on clinical evaluation,placebo-controlled infusion will be stopped 15 minutes before the end of surgery.Propofol and remifentanil infusion will be stopped at the end of surgery.
  Arms: sodium chloride (NaCl; 0.9%)
Drug: S-ketamine — For patients in the s-ketamine group,anaesthesia will be maintained with s-ketamine infusion（0.3mg/kg/h),while anaesthesia will be maintained with propofol infusion(4-12mg/kg/h),analgesia will be maintained with remifentanil(0.15-0.3ug/kg/min).The sufentanil dose at induction and the rate of intraoperative remifentanil and propofol infusions were at the discretion of the anesthesiologist in charge of the patient.The assessment of the depth of anesthesia was based on clinical evaluation.S-ketamine infusion will be stopped 15 minutes before the end of surgery.Propofol and remifentanil infusion will be stopped at the end of surgery.
  Arms: S-ketamine

SUMMARY:
Severe acute pain after total knee arthroplasty surgery has multiple implications for hospitals and patients, monopolising resources and affecting the quality of life. S-ketamine inhibits N-methyl-d-aspartate (NMDA) receptor activation and attenuates central sensitization associated with hyperalgesia, opioid tolerance.Therefore, the primary aim of this trial was to investigate whether s-ketamine decreases pain and opioid consumption postoperatively in adult individuals undergoing total knee arthroplasty surgery.

DETAILED DESCRIPTION:
Total knee arthroplasty surgery is considered a cost-effective therapy for end-stage knee osteoarthritis (KOA). With an ageing population and rising rates of obesity in the world, knee joint replacements are estimated to escalate. While joint replacement is a cost effective intervention,approximately 20% of people experience persist pain postoperatively. The surgical injury triggers a myriad of responses in the pain matrix, from sensitization of peripheral and central pain pathways to feelings of fear, anxiety and frustration.

Opioids are effective for acute postoperative pain but have numerous adverse effects. In addition, postoperative opioid treatment may pose a risk of opioid addiction.

Numerous publications state that adjuvant s-ketamine reduces pain and opioid consumption postoperatively . Whether intraoperative intravenous s-ketamine alleviates postoperative acute pain after total knee arthroplasty surgery still unclear . Therefore, a randomized, controlled, clinical study was designed to observed analgesic effect intraoperative intravenous a lower doses of s-ketamine(0.3mg/kg/h) with patients after total knee arthroplasty surgery .

ELIGIBILITY:
Inclusion Criteria:

1. ASA physical statusI-III;
2. Patients understood the study in detail and voluntarily signed the informed consent before the study;
3. Patients to be treated with total knee arthroplasty Surgery under General anesthesia;
4. Elderly patients(≥65y),regardless of gender;
5. Patients can communicate normally;
6. Patients who have no contraindications to drugs such as midazolam,fentanyl,s-ketamine.

7.18 kg/m2 ≤BMI≤30 kg/m2;

Exclusion Criteria:

1. Increased intracranial or intraocular pressure;
2. severe hypertension;
3. unwillingness the study;
4. severe psychiatric disease and mental system diseases;
5. severe respiratory diseases;
6. hyperthyroidism;
7. liver and kidney dysfunction;
8. alcohol or drug abuse;
9. allergy to midazolam,fentanyl,s-ketamine.

Ages: 65 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 144 (Estimated)
Dates: Start 2022-04-19 (Actual); Primary Completion 2024-09-01 (Estimated); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
at rest and movement, evaluated NRS at 24hours after surgery in the surgical ward. | the patient at 24hours after operation.
  NRS = (numerical rating scale) is widely used to measure pain intensity after surgery.NRS is evaluated on a 11-point NRS (0 = no pain, 10 = worst pain imaginable)

SECONDARY OUTCOMES:
at rest and movement, evaluated NRS at 2 hours after surgery in the surgical ward. | the patient at 2 hours after operation.
  NRS = (numerical rating scale) is widely used to measure pain intensity after surgery.NRS is evaluated on a 11-point NRS (0 = no pain, 10 = worst pain imaginable)
at rest and movement, evaluated NRS at 48hours after surgery in the surgical ward. | the patient at 48hours after operation
  NRS = (numerical rating scale) is widely used to measure pain intensity after surgery.NRS is evaluated on a 11-point NRS (0 = no pain, 10 = worst pain imaginable)
The cumulative Opioids consumption during the first 48h after operation | Within 48hours after surgery
  The cumulative Opioids consumption such as demerol,sufentanil,morphine
The number of patients who required additional analgesics during the first 48h after operation | Within 48hours after surgery
  The number of patients who required additional analgesics such as opioids(demerol,sufentanil,morphine)or non-steroid anti-inflammatory drugs(acetaminophen,diclofenac).
The Opioids or non-steroid anti-inflammatory drugs total consumption during the first 48h after operation | Within 48hours after surgery
  The opioids (such as demerol,sufentanil,morphine) or non-steroid anti-inflammatory drugs (such as acetaminophen,diclofenac)total consumption.
The incidence of PONV and adverse central nervous system (CNS) events. | at2, 24, 48hours after operation.
  (Postoperative nausea and vomiting)Nausea is defined as subjective,unpleasant sensation associated with awareness of the urge to vomit. Retching is defined as the laboured, spastic, rhythmic contraction of the respiratory muscles without expulsion of the gastric contents.Vomiting is defined as the forceful expulsion of gastric contents from the mouth.The adverse central nervous system (CNS) events(such as nightmares, hallucinations, dizziness, itchy skin) were recorded (yes/no) at the patient leaves the PACU and at 24, 48hours in the surgical ward.

CONTACTS AND LOCATIONS:
Locations (1):
- Qianfoshan Hospital, The First Hospital affiliated of Shandong First Medical University, Jinan, Shandong, China

REFERENCES:
- [Derived] Deng SY, Song X, Chen LN, Zhao F, Guo L. The Analgesic Effect of Low-Dose S(+)-Ketamine in Knee Joint Replacement: A Randomized Controlled Trial. J Pain Res. 2025 Nov 4;18:5815-5826. doi: 10.2147/JPR.S545997. eCollection 2025. PMID 41209744
- [Derived] Deng S, Chen L, Song X, Guo L, Zhao F, Liu J, Dong L. Analgesic Effect of Intraoperative Intravenous S(+)-Ketamine During Total Knee Arthroplasty Surgery: Study Protocol for a Randomized Controlled Clinical Trial. JMIR Res Protoc. 2023 Dec 8;12:e53063. doi: 10.2196/53063. PMID 38064260